CLINICAL TRIAL: NCT03140215
Title: Comparative Study of Baska & I-Gel for Spontaneously Ventilated Females During Minor Gynecological Procedures
Brief Title: Comparative Study of Baska & I-gel for Ventilation of Female Patients During Minor Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesrine El-Refai, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UTF-8
Record Dates: First submitted 2016-01-08; First posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Medical Device Complication
Keywords: Baska; seal pressure; I-Gel; Supraglottic airway device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baska Device ventilation group (Active Comparator): Device: laryngeal mask insertion (Baska)
  Interventions: Device: laryngeal mask insertion (Baska); Device: laryngeal mask insertion (I-gel )
- I-Gel device ventilation group (Active Comparator): Device: laryngeal mask insertion ( I-gel )
  Interventions: Device: laryngeal mask insertion (Baska); Device: laryngeal mask insertion (I-gel )

INTERVENTIONS:
Device: laryngeal mask insertion (Baska)
  Other Names: Baska
Device: laryngeal mask insertion (I-gel )
  Other Names: I-gel

SUMMARY:
The study aimed to compare safety of the 3rd generation Supra-glottic airway device (SAD) "Baska" to the I-Gel , regarding seal pressure, fitting on the larynx (detected by Fiberoptic) & complications. The study will be done for females undergoing minor gynecological procedures under general anesthesia with spontaneous ventilation.

DETAILED DESCRIPTION:
Population of study & disease condition : 2 equal groups (n=30), female patients enrolled for minor gynecological procedures (D&C or hysteroscopy), All patients received general anesthesia with spontaneous ventilation using Supra-glottic airway Device (SAD). Group A (Baska) & group B ( I-gel).

Inclusion Criteria: Age: 18-55, American Society of Anesthesia (ASA) 1 or 2, BMI<35 & Low risk of aspiration.

Exclusion Criteria: Anticipated upper airway problem, Gastrointestinal tract (GIT, disease, pregnancy & High risk of aspiration.

Methodology: All patients received fentanyl 1 micro gram/Kg, Propofol(2-4mg/Kg) was titrated to induce anesthesia, followed by manual ventilation with sevoflurane (2-4%) in Oxygen.All devices were inserted by one of 2 investigators.

Data collection: 1- Demographic Data: age,weight,height.2-duration of anesthesia.3- Data related to device insertion: Time of insertion,duration of anesthesia, seal pressure,peak airway pressure, Fiberoptic (FO)view of the larynx ,vomiting or regurgitation, postoperative laryngeal spasm or blood on the device after removal.

Primary outcome: To detect seal pressure and fitting against laryngeal aperture detected by FO. Secondary outcome:To determine Peak pressure, incidence of complications: vomiting or regurgitation, blood on the device after removal (indicating trauma to the airway) or postoperative laryngeal spasm..

Statistical analysis: For analysis of continuous variables independent sample t-test will be applied and for categorical variables chi-square test will be used.value of p<0.05 will be considered significant.

Sample size:

Sample size was calculated using EpiCalc program using the following data : mean seal pressure for Baska :29.98 , mean seal pressure for I-Gel: 25.62. SD: 4.9

, study power 80% confidence interval . P value<0.05. the calculated sample size was found to be 19 for each group (overall 38), so the investigators will allocate 30 patient in each group to avoid drop out.

Statistical analysis:

Source of funding This study will be attributed to Department of Anesthesiology, Faculty of medicine, Cairo University. Support will be provided solely from departmental sources. Keywords: Baska, I-Gel, Supra-glottic airway devices, seal pressure

ELIGIBILITY:
Inclusion Criteria:

* Female ASA1,2
* Age 18-55
* BMI<35

Exclusion Criteria:

* Anticipated upper airway problem
* GIT disease
* Pregnancy
* High risk of aspiration

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
seal pressure | seal pressure will be assessed 3minutes after induction of general anesthesia.
  Airway Sealing Pressure in cmH2O at 5 mins postplacement.The airway sealing pressure was the pressure at which leak starts. This leak pressure was calculated as the plateau airway pressure reached with fresh gas flow 6 l/min, and pressure adjustment valve set at 70 cmH2O..

SECONDARY OUTCOMES:
Fiberoptic view of the larynx. | Fiberoptic view will be assessed 5 minutes after induction of anesthesia.
  The fiberoptic device will be introduced through the device to visualize & record the view
Peak airway pressure in CmH2O | during the operation the operation
  The peak airway pressure will be monitored during the operation time
incidence of vomiting and regurgitation | from the start of operation till 10 minutes postoperative
  patients will be monitored to detect vomiting & regurgitation.

CONTACTS AND LOCATIONS:
Overall Officials: Nesrine A. El-Refai, M.D, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided